CLINICAL TRIAL: NCT02008318
Title: Phase 2/3 Study of Monotherapy LY2157299 Monohydrate in Very Low-, Low-, and Intermediate-Risk Patients With Myelodysplastic Syndromes
Brief Title: A Study of Galunisertib in Participants With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15242; H9H-MC-JBAV (Other: Eli Lilly and Company); 2013-003235-30 (EudraCT Number)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — LY-2157299

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase (ph) 2: Galunisertib + BSC (Experimental): Ph 2. 150 milligrams Galunisertib given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles). Participants will receive best supportive care (BSC) according to institutional guidelines. Treatment is expected to last for 6 cycles. Participants may receive additional cycles if they are deriving clinical benefit.
  Interventions: Drug: Galunisertib
- Ph 3: Placebo + BSC (Placebo Comparator): Placebo administered orally BID for 14 days followed by 14 days with no study drug (28 day cycles). Participants will receive BSC according to institutional guidelines. Treatment is expected to last for 6 cycles. Participants may receive additional cycles if they are deriving clinical benefit. This arm is contingent on the data from the phase 2 arm.
  Interventions: Drug: Placebo
- Ph 3: Galunisertib + BSC (Experimental): 150 milligrams Galunisertib given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles). Participants will receive best supportive care (BSC) according to institutional guidelines. Treatment is expected to last for 6 cycles. Participants may receive additional cycles if they are deriving clinical benefit. This arm is contingent on the data from the phase 2 arm.
  Interventions: Drug: Galunisertib

INTERVENTIONS:
Drug: Galunisertib — Administered orally
  Other Names: LY2157299
  Arms: Ph 3: Galunisertib + BSC; Phase (ph) 2: Galunisertib + BSC
Drug: Placebo — Administered orally
  Arms: Ph 3: Placebo + BSC

SUMMARY:
The purpose of this study is to investigate the effect of the study drug known as galunisertib in participants with myelodysplastic syndromes (MDS). Participants with different degrees of disease (very low, low, and intermediate risk) will be studied. The study treatment is expected to last about 6 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MDS based on the World Health Organization (WHO) criteria
* Participants with 5q deletions are allowed only if they have failed or are intolerant of lenalidomide treatment
* Participants must have a Revised International Prognostic Scoring System (IPSS-R) category of very low-, low-, or intermediate-risk disease
* In the 8 weeks prior to registration, participants in phase 2 should have anemia with Hb ≤10.0 g/dL (based on the average of 2 baseline measurements and untransfused for at least 1 week) with or without red blood cell (RBC) transfusion dependence confirmed for a minimum of 8 weeks before enrollment
* For phase 3, participants should have anemia with RBC transfusion dependence confirmed within 8 weeks before enrollment
* Performance status ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale

Exclusion Criteria:

* No history of moderate or severe cardiac disease
* No prior history of acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westerstede
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Santini V, Valcarcel D, Platzbecker U, Komrokji RS, Cleverly AL, Lahn MM, Janssen J, Zhao Y, Chiang A, Giagounidis A, Guba SC, Gueorguieva I, Girvan AC, da Silva Ferreira M, Bhagat TD, Pradhan K, Steidl U, Sridharan A, Will B, Verma A. Phase II Study of the ALK5 Inhibitor Galunisertib in Very Low-, Low-, and Intermediate-Risk Myelodysplastic Syndromes. Clin Cancer Res. 2019 Dec 1;25(23):6976-6985. doi: 10.1158/1078-0432.CCR-19-1338. Epub 2019 Sep 3. PMID 31481511

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single-arm study (Galunisertib at 150 milligram [mg]); the Galunisertib at 80 mg was considered exploratory and only conducted in parallel with the main study, at one site in Spain.
Groups:
- Galunisertib at 150 mg: Galunisertib at 150 mg given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles).
- Galunisertib at 80 mg: Exploratory arm: Galunisertib at 80 mg given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles).
Period: Overall Study
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Started | 41 | 2
Received At Least 1 Dose of Study Drug | 41 | 2
Completed (Completed at least 6 cycles) | 29 | 1
Not Completed | 12 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Progressive Disease | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants (including the Galunisertib at 80 mg exploratory arm) who received at least one dose of study drug.
Groups:
- Galunisertib at 150 mg: Galunisertib at 150 mg given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles). Participants will receive best supportive care (BSC) according to institutional guidelines.
- Galunisertib at 80 mg: Exploratory arm: Galunisertib at 80 mg given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles). Participants will receive best supportive care (BSC) according to institutional guidelines.
- Total: Total of all reporting groups
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg | Total
Number analyzed (Participants) | 41 | 2 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.49 (7.65) | 62.50 (10.61) | 70.12 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 1 | 16
  Male | 26 | 1 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 32 | 2 | 34
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 2 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 8 | 0 | 8
  Germany | 23 | 0 | 23
  Spain | 10 | 2 | 12
IPSS-R Prognostic Risk Score [Count of Participants; unit: Participants] — Revised International Prognostic Scoring System (IPSS-R) is a screening tool used for MDS risk assessment. IPSS-R gives great weight to cytogenetic abnormalities and severity of cytopaenias, while reassigning the weighting for blast percentages.
  Score Categories: ≤1.5 Very Low, >1.5 - 3 Low, >3 - 4.5 Intermediate, >4.5 - 6 High, >6 Very High.
  The MDS Foundation website provides a calculator for determining IPSS-R scoring.
  Participants
    Very Low= (≤1.5) | 2 | 0 | 2
    Low= (>1.5 - 3) | 30 | 1 | 31
    Intermediate= (>3 - 4.5) | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hematological Improvement (HI)
Description: Percentage of participants with hematological improvement (HI) based on International Working Group (IWG) 2006 criteria in participants with very low, low, and intermediate-risk myelodysplastic syndromes treated with Galunisertib plus best supportive care, as assessed by the International Prognostic Scoring System (IPSS-R).
  To be classified as an HI responder, the HI response must have lasted at least 8 weeks (56 days).
Time Frame: Baseline through end of study treatment (24 weeks)
Population: Participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm: Galunisertib at 80 mg: Exploratory arm: Galunisertib at 80 mg given orally twice daily (BID) for 14 days followed by 14... more days with no study drug (28 day cycles). Completed participants completed at least 6 cycles.
Arm/Group | Galunisertib at 150 mg | Arm: Galunisertib at 80 mg
Number analyzed (Participants) | 41 | 2
percentage of participants | 31.7 [18.1 to 48.1] | 0.0 [0.0 to 84.2]

2. Primary Outcome: Percentage of Participants Who Are Transfusion-free or Have Hemoglobin (Hb) Increase ≥1.5 Grams/Deciliter Maintained for 8 Weeks During Phase 3
Description: Comparison of the percentage of participants with very low-, low-,and intermediate-risk MDS who were transfusion-free or had an increase ≥1.5 g/dL in hemoglobin (Hb) maintained for at least 8 weeks within the first 24 weeks of treatment with galunisertib plus best supportive care or placebo plus best supportive care and assessed by IPSS-R.
  The Phase 3 portion of this study was not conducted because efficacy level required in phase 2 to move forward to phase 3 was not achieved.
Time Frame: Baseline through end of study treatment (24 weeks)
Population: Participants who received at least one dose of study drug during Phase 3.
Groups:
- Galunisertib at 80 mg: Exploratory arm: Galunisertib at 80 mg given orally twice daily (BID) for 14 days followed by 14... more days with no study drug (28 day cycles). Completed participants completed at least 6 cycles.
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI)
Description: The Brief Fatigue Inventory (BFI) is a brief participant-reported questionnaire that measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours. The severity of fatigue is assessed using an 11-point numeric scale, with 0 = no fatigue and 10 = fatigue as bad as you can imagine.
Time Frame: Baseline, Follow up (final visit up to 24 months)
Population: Participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Number analyzed (Participants) | 41 | 2
units on a scale
  Current Fatigue at Follow-up | 0.818 (0.42) | -1.005 (2.08)
  Usual Fatigue at Follow-up | -0.017 (0.37) | -0.157 (1.87)
  Worst Fatigue at Follow-up | -0.191 (0.38) | -0.063 (1.93)

4. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 5 Level Instrument
Description: EuroQol 5-Dimension 5 Level Instrument (EQ-5D-5L) was not conducted, trial terminated prior to Phase 3. No data collected.
Time Frame: Phase 3: Baseline, Cycle 2, Cycle 4, Cycle 6 (Cycle = 28 days)
Population: Participants who received at least one dose of study drug during Phase 3.
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Cytogenetic Response
Description: Percentage of Participants with Cytogenetic Response with either complete or partial response. Complete cytogenetic response is the disappearance of the chromosomal abnormality without appearance of new ones. Partial cytogenetic response is at least 50% reduction of the chromosomal abnormality.
Time Frame: Baseline through end of study treatment (24 weeks)
Population: Participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Number analyzed (Participants) | 41 | 2
percentage of participants | 2.4 [0.1 to 12.9] | 0 [0 to 0]

6. Secondary Outcome: Percentage of Participants Who Are Hospitalized (Resource Utilization)
Description: Percentage of any participant with a hospitalization admission and discharge date on the same day are counted as a half-day in the duration of hospitalization.
Time Frame: Baseline through end of study treatment (24 weeks)
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Number analyzed (Participants) | 41 | 2
percentage of participants | 24.3 | 0

7. Secondary Outcome: Population Pharmacokinetics (PK): Mean Population Clearance of Galunisertib
Description: Population mean (between-participant coefficient variation [CV%]) apparent clearance.
Time Frame: Day 1 pre-dose & between 0.5 to 2 hours post dose; Day 14 pre-dose, between 0.5 to 2 & between 3 to 5 hours post dose; Days 15 & 16 (if logistically possible) between 0.5 to 2 hours post dose
Population: All participants who received at least one dose of study drug, regardless of dose, with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Groups:
- Galunisertib: Galunisertib given orally twice daily (BID) for 14 days followed by 14 days with no study drug (28 day cycles).
Arm/Group | Galunisertib
Number analyzed (Participants) | 43
Liter per hour (L/h) | 32 (52)

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of first dose to the date of death from any cause.
Time Frame: Baseline to date of death from any cause (Up to 2 years)
Population: Participants who received at least one dose of study drug excluding the exploratory participants.
Measure: Median (Full Range); unit: days
Arm/Group | Galunisertib at 150 mg
Number analyzed (Participants) | 41
days | 679 [29 to 729]

9. Secondary Outcome: Number of Participants With a Change in Bone Marrow Fibrosis Grading
Description: Change from baseline in bone marrow fibrosis measured the number of participants with a change in bone marrow fibrosis grading (negative, mild, moderate, and severe).
Time Frame: Baseline, Cycle 6 (Cycle = 28 days)
Population: Participants who received at least one dose of study drug and had both a baseline and postbaseline assessment excluding the exploratory participants.
Measure: Number; unit: participants
Arm/Group | Galunisertib at 150 mg
Number analyzed (Participants) | 30
participants | 11

ADVERSE EVENTS:
Time Frame: Baseline through end of study treatment or death from any cause (Up to 2 years)
Arm/Group | Galunisertib at 150 mg | Galunisertib at 80 mg
Serious Adverse Events (participants affected / at risk) | 8/41 | 0/2
Other Adverse Events (participants affected / at risk) | 33/41 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galunisertib at 150 mg (N=41) | Galunisertib at 80 mg (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Tongue abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galunisertib at 150 mg (N=41) | Galunisertib at 80 mg (N=2)
Anaemia (Blood and lymphatic system disorders) | 3 (18) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0)
Asthenia (General disorders) | 5 (13) | 1 (1)
Fatigue (General disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 5 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The response rate at interim analysis did not meet the predefined rate. The Phase 3 portion was not initiated and the sponsor decided on early discontinuation of the study at the conclusion of Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days